CLINICAL TRIAL: NCT06066203
Title: An Open, Multicenter, Phase I / II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics / Pharmacodynamics and Antitumor Activity of GNC-035 Tetra-specific Antibody Injection in Relapsed or Refractory Non-Hodgkin 's Lymphoma and Other Hematological Malignancies
Brief Title: A Study of GNC-035 in Relapsed or Refractory Non-Hodgkin 's Lymphoma and Other Hematological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-035-104
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Non-hodgkin's Lymphoma
Keywords: Hematological malignancies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-035 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-035

INTERVENTIONS:
Drug: GNC-035 — GNC-035 was administered by intravenous infusion for 2 h-4 h, once a week ( IV, QW ), 3 weeks as a cycle.

SUMMARY:
Phase I main objectives: To observe the safety and preliminary efficacy of GNC-035 in patients with relapsed/refractory non-Hodgkin lymphoma and other hematological malignancies, to determine the DLT and MTD, or MAD, and to determine RP2D. Phase II Main objective: To explore the efficacy of GNC-035 in patients with relapsed/refractory non-Hodgkin lymphoma and other hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to understand the informed consent form, voluntarily participates, and signs the informed consent form;
2. No gender restrictions;
3. Age: ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Histologically or cytologically confirmed relapsed or refractory non-Hodgkin's lymphoma;
6. For patients with relapsed or refractory non-Hodgkin's lymphoma, specifically including: Patients who have failed at least one line of standard therapy; Patients with relapsed or refractory disease judged by the investigator to have no other available or suitable treatment options;
7. For non-Hodgkin's lymphoma, at least one measurable lesion meeting the Lugano response criteria must be present during the screening period;
8. ECOG performance status score ≤2;
9. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. Organ function levels meet the requirements within 7 days before the first dose;
11. Female subjects of childbearing potential or male subjects with partners of childbearing potential must use highly effective contraception from 7 days before the first dose until 12 weeks after the last dose. Female subjects of childbearing potential must have a negative serum/urine pregnancy test within 7 days before the first dose;
12. The subject has the ability and willingness to comply with the study protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Patients who have undergone major surgery within 28 days prior to the administration of this study or are scheduled for major surgery during the study period (major surgery is defined by the investigator);
2. Pulmonary diseases classified as ≥Grade 3 according to NCI-CTCAE v5.0;
3. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
4. Patients with active autoimmune diseases;
5. History of other malignancies within 5 years prior to the first dose;
6. Positive for human immunodeficiency virus (HIV) antibodies, active tuberculosis, active hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection;
7. Poorly controlled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg) despite medication;
8. History of severe cardiovascular or cerebrovascular diseases;
9. Patients with a history of hypersensitivity to recombinant humanized antibodies or any excipients of GNC-035;
10. Pregnant or lactating women;
11. Patients with central nervous system involvement;
12. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
13. Autologous hematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks before initiating GNC-035 treatment;
14. Current use of immunosuppressive therapy;
15. Radiotherapy or macromolecular targeted therapy within 4 weeks before initiating GNC-035 treatment; chemotherapy or small-molecule targeted therapy within 2 weeks or 5 half-lives (whichever is shorter) before treatment;
16. Anti-CD20 or anti-CD79b treatment within 4 weeks before initiating GNC-035 treatment with ongoing response;
17. CAR-T therapy within 12 weeks before initiating GNC-035 treatment;
18. Use of investigational drugs from other clinical trials within 4 weeks or 5 half-lives (whichever is shorter) before the administration of this study;
19. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase I: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase I: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-035. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-035.
Phase I: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-035.
Phase II: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase I: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-035 to the first date of either disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase I: Complete Response (CR) | Up to approximately 24 months
  Complete response (CR) is defined as all tumor target lesions disappeared, no new lesions appeared, and tumor markers were normal for at least 4 weeks.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-035. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-035.
Phase I: Cmax | Up to 21 days after the first dose
  Maximum Drug Concentration (Cmax) of GNC-035 will be investigated.
Phase I: Tmax | Up to 21 days after the first dose
  Time at Which the Maximum (Tmax) of GNC-035 will be investigated.
Phase I: AUC0-inf | Up to 21 days after the first dose
  Area Under the Curve（0-inf）of GNC-035 will be investigated.
Phase I: AUC0-T | Up to 21 days after the first dose
  Area Under the Curve（0-t）of GNC-035 will be investigated.
Phase I: CL | Up to 21 days after the first dose
  Rate of clearance of GNC-035 will be investigated.
Phase Ib: T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of GNC-035 will be investigated.
Phase I: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-GNC-035 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China